CLINICAL TRIAL: NCT00824889
Title: Exploratory Study of Natural Killer Cells in Human Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2008-A00064-51; 2008-03
Record Dates: First submitted 2009-01-13; First posted 2009-01-19 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Atopic Dermatitis; Contact Dermatitis; Psoriasis; Lichen Planus; Graft Versus Host Disease; Melanoma
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis, Contact; Psoriasis; Lichen Planus; Graft vs Host Disease; Melanoma | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Other): Healthy volunteer
  Interventions: Other: Biopsy and sample of blood
- 2 (Other): atopic dermatitis patient
  Interventions: Other: Biopsy and sample of blood
- 3 (Other): contact dermatitis patient
  Interventions: Other: Biopsy and sample of blood
- 4 (Other): psoriasis patient
  Interventions: Other: Biopsy and sample of blood
- 5 (Other): lichen planus patient
  Interventions: Other: Biopsy and sample of blood
- 6 (Other): GVH patient
  Interventions: Other: Biopsy and sample of blood
- 7 (Other): melanoma patient
  Interventions: Other: Biopsy and sample of blood

INTERVENTIONS:
Other: Biopsy and sample of blood — Biopsy and sample of blood
  Arms: 1
Other: Biopsy and sample of blood — Biopsy and sample of blood
  Arms: 2
Other: Biopsy and sample of blood — Biopsy and sample of blood
  Arms: 3
Other: Biopsy and sample of blood — Biopsy and sample of blood
  Arms: 4
Other: Biopsy and sample of blood — Biopsy and sample of blood
  Arms: 5
Other: Biopsy and sample of blood — Biopsy and sample of blood
  Arms: 6
Other: Biopsy and sample of blood — Biopsy and sample of blood
  Arms: 7

SUMMARY:
Natural Killer (NK) cells play a unique role during innate immune responses as they are able to recognize and eliminate, without specific sensitization, tumors, microbe-infected cells as well as allogeneic cells.In a first time, we will characterize the tissue distribution, the phenotype and the effector functions of NK cells present in the human healthy skin.

DETAILED DESCRIPTION:
Then, we will define whether these parameters are qualitatively/ quantitatively modified in the following skin pathologies: a) atopic dermatitis; b) contact dermatitis; c) psoriasis ; d) lichen planus ; e) GVH (graft versus host disease) ; (f) melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Consent obtained after healthy donor or patient information.
* Patients suffering from one of the following diseases: a) atopic dermatitis ; b) contact dermatitis; c) psoriasis ; d) lichen planus ; e) GVH ; f) melanoma.

Exclusion Criteria:

* Age below 18,
* pregnant or breastfeeding women,
* persons under guardianship, persons without social security, prisoners, persons hospitalized without consent on the basis of French laws L. 3212-1 et L. 3213-1. Patients affected by HIV infection, AIDS, Hepatitis A, B or C infection.
* Neutropenia <1000/mm3.
* Thrombopenia <50 000/mm3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
In a first time, we will characterize the tissue distribution, the phenotype and the effector functions of NK cells present in the human healthy skin. | 12 months

SECONDARY OUTCOMES:
To determine whether the eventual modifications detected in skin pathologies are correlated to qualitative/ quantitative alterations of NK cell subsets present in the peripheral blood. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Gaudy-Marqueste, MD, Principal Investigator — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Service de Dermatologie- Hopital Sainte Marguerite, Marseille, France